CLINICAL TRIAL: NCT03496207
Title: A Phase 2, Double-Blind, Placebo-Controlled, Randomized Study to Compare the Efficacy and Safety of Sotatercept (ACE-011) Versus Placebo When Added to Standard of Care for the Treatment of Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study of Sotatercept for the Treatment of Pulmonary Arterial Hypertension (PAH)
Acronym: PULSAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A011-09; 2017-004738-27 (EudraCT Number)
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — ACE-011

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo plus SOC by SC injection during the 24-week treatment period. Dosing will occur once every 3 weeks.
  Interventions: Drug: Placebo; Other: SOC
- Sotatercept 0.3 mg/kg (Experimental): Participants will receive sotatercept 0.3 mg/kg plus SOC by SC injection during the 24-week treatment period. Per protocol, participants may have their doses titrated. Dosing will occur once every 3 weeks.
  Interventions: Drug: Sotatercept; Other: SOC
- Sotatercept 0.7 mg/kg (Experimental): Participants will receive sotatercept 0.7 mg/kg plus SOC by SC injection during the 24-week treatment period. Per protocol, participants may have their doses titrated. Dosing will occur once every 3 weeks.
  Interventions: Drug: Sotatercept; Other: SOC

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Sotatercept — Sotatercept (ACE-011) is a recombinant fusion protein consisting of the extracellular domain of the human activin receptor type IIA linked to the Fc piece of human IgG1.
  Other Names: ACE-011
  Arms: Sotatercept 0.3 mg/kg; Sotatercept 0.7 mg/kg
Other: SOC — SOC therapy refers to approved PAH-specific medications and may consist of monotherapy or combination therapy with endothelin-receptor antagonists, phosphodiesterase 5 (PDE5) inhibitors, soluble guanylate cyclase stimulators, and/or prostacyclin analogues or receptor agonists.

SUMMARY:
Study A011-09 is designed to assesses the efficacy and safety of sotatercept (ACE-011) relative to placebo in adults with pulmonary arterial hypertension (PAH). Eligible participants will receive study treatment for 24 weeks during the placebo-controlled treatment period, and then will be eligible to enroll into a 30-month extension period during which all participants will receive sotatercept. All treated patients will also undergo a follow-up period after last study drug treatment.

DETAILED DESCRIPTION:
This is a Phase 2, double-blind, randomized, placebo-controlled, parallel-group study of sotatercept plus standard of care (SOC) versus placebo plus SOC in participants with PAH of World Health Organization (WHO) Group 1, functional class II-III. Participants will be randomly assigned in a 3:3:4 ratio to receive placebo, sotatercept 0.3 mg/kg, or sotatercept 0.7 mg/kg by subcutaneous (SC) injection every 21 days for a period of 24 weeks in the placebo-controlled treatment period of the study while on SOC therapy. Evaluations will include changes in pulmonary vascular resistance (PVR), 6-minute walk distance (6MWD), quality of life questionnaires, echocardiographic parameters, and safety. Participants who have not discontinued early from the placebo-controlled treatment period and have had their post-treatment period PVR assessment will be able to continue into the 30-month extension period in which sotatercept-treated participants will receive their latest dose level of sotatercept SC every 21 days and placebo-treated participants will be re-randomized 1:1 to receive sotatercept 0.3 mg/kg SC or sotatercept 0.7 mg/kg SC every 21 days while on SOC therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Documented diagnostic right heart catheterization (RHC) at any time prior to Screening confirming diagnosis of WHO diagnostic pulmonary hypertension Group I: PAH in any of the following subtypes:

   i. Idiopathic ii. Heritable PAH iii. Drug- or toxin-induced PAH iv. PAH associated with connective tissue disease v. PAH associated with simple, congenital systemic-to-pulmonary shunts at least 1 year following shunt repair
3. Symptomatic pulmonary hypertension classified as WHO functional class II or III
4. Screening RHC documenting a minimum PVR of ≥400 dyn·sec/cm5 (5 Wood units)
5. Pulmonary function tests (PFTs) within 6 months prior to Screening as follows:

   1. Total lung capacity (TLC) >70% predicted; or if between 60 to 70% predicted, or not possible to be determined, confirmatory high-resolution computed tomography (CT) indicating no more than mild interstitial lung disease (ILD), per investigator interpretation, or
   2. Forced expiratory volume (first second) (FEV1)/ forced vital capacity (FVC) >70% predicted
6. Ventilation-perfusion (VQ) scan (or, if unavailable a negative CT pulmonary angiogram [CTPA] result, or pulmonary angiography result), any time prior to Screening Visit or conducted during the Screening Period, with normal or low probability result),
7. No contraindication per investigator for RHC during the study
8. 6MWD ≥150 and ≤550 meters repeated twice at Screening and both values within 15% of each other, calculated from the highest value
9. PAH therapy at stable (per investigator) dose levels of SOC therapies

Exclusion Criteria:

1. Stopped receiving any pulmonary hypertension chronic general supportive therapy (e.g, diuretics, oxygen, anticoagulants, digoxin) within 60 days prior to study visit Cycle 1 Day 1 (C1D1)
2. Received intravenous inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to study visit C1D1
3. History of atrial septostomy within 180 days prior to Screening
4. History of more than mild obstructive sleep apnea that is untreated
5. Known history of portal hypertension or chronic liver disease, including hepatitis B and/or hepatitis C (with evidence of recent infection and/or active virus replication), defined as mild to severe hepatic impairment (Child-Pugh Class A-C)
6. History of human immunodeficiency virus infection-associated PAH
7. Prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536)
8. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to C1D1 or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible).
9. Uncontrolled systemic hypertension as evidenced by sitting systolic blood pressure (BP) >160 mm Hg or sitting diastolic blood pressure >100 mm Hg during Screening Visit after a period of rest
10. Systolic BP <90 mmHg during Screening or at baseline
11. History of known pericardial constriction
12. Electrocardiogram (ECG) with Fridericia's corrected QT interval (QTcF) >480 msec during Screening Period or C1D1
13. Personal or family history of long QTc syndrome or sudden cardiac death
14. Cerebrovascular accident within 3 months of C1D1
15. History of restrictive or congestive cardiomyopathy
16. Left ventricular ejection fraction (LVEF) <45% on historical echocardiogram (ECHO) within 6 months prior to Screening Period (or done as a part of the Screening Period) or pulmonary capillary wedge pressure (PCWP) >15 mmHg as determined in the Screening Period RHC.
17. Any current or prior history of symptomatic coronary disease (prior myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain)
18. Acutely decompensated heart failure within 30 days prior to study visit C1D1, as per investigator assessment
19. Significant (≥2+ regurgitation) mitral regurgitation (MR) or aortic regurgitation (AR) valvular disease
20. Any of the following clinical laboratory values during the Screening Period prior to C1D1:

    1. Baseline Hgb >16.0 g/dL
    2. Serum alanine aminotransferase or aspartate aminotransferase levels >3X upper limit of normal (ULN) or total bilirubin >1.5X ULN within 28 days of C1D1
    3. Estimated glomerular filtration rate <30 ml/min/1.73m2 (4-variable Modification of Diet in Renal Disease equation) within 28 days of C1D1 or required renal replacement therapy within 90 days
    4. WBC count <4000/mm3
    5. Platelets <100,000/μL
    6. Absolute neutrophil count <1500/mm3
21. History of opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia) within 6 months prior to Screening; serious local infection (e.g., cellulitis, abscess) or systemic infection (e.g., septicemia) within 3 months prior to Screening
22. History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients in the investigational product
23. Major surgery within 8 weeks prior to C1D1. Participants must have completely recovered from any previous surgery prior to C1D1.
24. Prior heart or heart-lung transplants or life expectancy of <12 month
25. Pregnant or breastfeeding females
26. If on corticosteroids, and at any time in the last 30 days prior to the Screening Period: have been receiving doses of >20 mg/day of prednisone (or equivalent) or on a new or changing dose of ≤20 mg/day; only participants receiving stable doses of ≤20 mg prednisone (or equivalent) in last 30 days prior to the Screening Period permitted in the study
27. History of active malignancy, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤2 squamous cell carcinomas of the skin
28. History of clinically significant (as determined by the investigator) non-PAH related cardiac, endocrine, hematologic, hepatic, (auto)immune, metabolic, urologic, pulmonary, neurologic, neuromuscular, dermatologic, psychiatric, renal, and/or another disease that may limit participation in the study. Autoimmune diseases are excluded with the exception of those related to PAH etiologies included in this study.
29. Participation in another clinical trial involving intervention with another investigational drug, approved therapy for investigational use, or investigational device within 4 weeks prior to C1D1, or if the half-life of the previous product is known, within 5 times the half-life prior to C1D1, whichever is longer
30. Weight >140 kg at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (43):
- United States (12):
  - Pulmonary Associates, PA, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Phoenix, Arizona
  - Banner-University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - University of California, San Francisco Medical Center, San Francisco, California
  - University of Colorado Hospital, Aurora, Colorado
  - UF Health Shands Hospital, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Lindner Clinical Trial Center, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Hospital, Houston, Texas
- Australia (4):
  - St. Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - John Hunter Hospital, New Lambton, New South Whales
  - Prince Charles Hospital, Chermside, Queensland
- Brazil (6):
  - Hospital Madre Teresa, Belo Horizonte, Minas Gerais
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Riogrande Do Sul
  - Hospital Dia do Pulmão, Blumenau, Santa Catarina
  - Instituto do Coracao - HCFMUSP, Cerqueira César
  - Hospital Sao Lucas da PUCRS, Jardim Botânico
  - Hospital São Paulo, São Paulo
- France (4):
  - Hôpital Arnaud de Villeneuve, Montpellier, Hérault
  - CHU Michallon, La Tronche
  - Centre Hospitalier Universitaire de Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire de Saint Etienne, Saint-Etienne
- Germany (4):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitatsklinikum Leipzig, Leipzig, Saxony
  - Universitatsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden
- Israel (5):
  - Barzilai Medical Center, Ashkelon
  - Lady Davis Carmel Medical Center, Haifa
  - Meir Medical Center, Kefar Sava
  - Rabin Medical Center - PPDS, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
- Spain (5):
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (3):
  - Golden Jubilee National Hospital - PPDS, Clydebank
  - Royal Free London NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Humbert M, McLaughlin V, Gibbs JSR, Gomberg-Maitland M, Hoeper MM, Preston IR, Souza R, Waxman AB, Ghofrani HA, Escribano Subias P, Feldman J, Meyer G, Montani D, Olsson KM, Manimaran S, de Oliveira Pena J, Badesch DB. Sotatercept for the treatment of pulmonary arterial hypertension: PULSAR open-label extension. Eur Respir J. 2023 Jan 6;61(1):2201347. doi: 10.1183/13993003.01347-2022. Print 2023 Jan. PMID 36041750
- [Derived] Humbert M, McLaughlin V, Gibbs JSR, Gomberg-Maitland M, Hoeper MM, Preston IR, Souza R, Waxman A, Escribano Subias P, Feldman J, Meyer G, Montani D, Olsson KM, Manimaran S, Barnes J, Linde PG, de Oliveira Pena J, Badesch DB; PULSAR Trial Investigators. Sotatercept for the Treatment of Pulmonary Arterial Hypertension. N Engl J Med. 2021 Apr 1;384(13):1204-1215. doi: 10.1056/NEJMoa2024277. PMID 33789009

RESULTS

PARTICIPANT FLOW:
Groups:
- Extension Period: Placebo→Sotatercept 0.3 mg/kg: This treatment group represents participants from the Placebo arm who received placebo plus standard of care (SOC) by subcutaneous (SC) injection during the 24-week treatment period (Base Study; Cycles 1-8), then transitioned to the 30-month extension period (Cycles 9-51), during which they received sotatercept 0.3 mg/kg plus SOC by SC injection. Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Extension Period: Placebo→Sotatercept 0.7 mg/kg: This treatment group represents participants from the Placebo arm who received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8), then transitioned to the 30-month extension period (Cycles 9-51), during which they received sotatercept 0.7 mg/kg plus SOC by SC injection. Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Placebo: Participants received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Sotatercept 0.3 mg/kg: Participants received sotatercept 0.3 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) and 30-month extension period (Cycles 9-51). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Sotatercept 0.7 mg/kg: Participants received sotatercept 0.7 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) and 30-month extension period (Cycles 9-51). Each cycle was 21 days. Dosing occurred once every 3 weeks.
Period: Base Study
Arm/Group | Extension Period: Placebo→Sotatercept 0.3 mg/kg | Extension Period: Placebo→Sotatercept 0.7 mg/kg | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Started | 0 | 0 | 32 | 32 | 42
Completed | 0 | 0 | 30 | 31 | 36
Not Completed | 0 | 0 | 2 | 1 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 1
Period: Extension Period
Arm/Group | Extension Period: Placebo→Sotatercept 0.3 mg/kg | Extension Period: Placebo→Sotatercept 0.7 mg/kg | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Started | 15 | 15 | 0 | 31 | 36
Completed | 13 | 15 | 0 | 28 | 31
Not Completed | 2 | 0 | 0 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1
Not completed — Death | 1 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1 | 1
Not completed — Elevated hemoglobin levels | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg | Total
Number analyzed (Participants) | 32 | 32 | 42 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.6 (13.38) | 49.1 (14.34) | 49.8 (15.05) | 48.3 (14.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 29 | 37 | 92
  Male | 6 | 3 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 9 | 13 | 32
  Not Hispanic or Latino | 21 | 19 | 28 | 68
  Unknown or Not Reported | 1 | 4 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 3 | 4
  White | 30 | 31 | 37 | 98
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Change From Baseline in Pulmonary Vascular Resistance (PVR) at 24 Weeks
Description: Each participant's PVR, at resting supine, was measured by right heart catheterization at baseline and at 24 weeks.
Time Frame: Baseline and 24 weeks
Population: All randomized participants administered their assigned treatment who received at least 6 of the same doses during Base Study, had baseline and post-Base Study PVR assessment and End of Treatment (EOT) assessment. Note: Data from participants whose dose was down-titrated were analyzed according to dose received at least 6 times rather than dose originally assigned. Per protocol, only participants who consistently received in 0.3 mg/kg or 0.7 mg/kg of sotatercept were planned to be analyzed.
Measure: Mean (Standard Deviation); unit: dynes*sec/cm^5
Groups:
- Sotatercept 0.3 mg/kg: Participants received sotatercept 0.3 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Sotatercept 0.7 mg/kg: Participants received sotatercept 0.7 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 27 | 30
dynes*sec/cm^5
  Base Study: Change from Baseline in PVR at 24 Weeks | -27.6 (251.08) | -168.4 (262.93) | -258.9 (169.42)
  Baseline | 802.0 (331.05) | 772.0 (285.62) | 715.5 (267.11)
Statistical Analysis 1: Comparison: Placebo vs Sotatercept 0.3 mg/kg; Analysis based on calculated LS means; Test type: Superiority; p = 0.0030, ANCOVA; ANCOVA was used to compare change from baseline values with randomization stratification factor (WHO functional class) and baseline PVR as covariate; Difference in Least Squares Means = -151.1, 95% CI 2-sided [-249.59 to -52.63], Standard Error of Mean 49.53
Statistical Analysis 2: Comparison: Placebo vs Sotatercept 0.7 mg/kg; Analysis based on calculated LS means; Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -269.4, 95% CI 2-sided [-365.81 to -173.03], Standard Error of Mean 48.48

2. Primary Outcome: Extension Period: Change From Baseline in PVR (Delayed-Start Analysis)
Description: Each participant's PVR, at resting supine, was measured by right heart catheterization at baseline and the timepoint at which the third right heart catheterization was performed, which occurred between Month 18 and Month 24.
Time Frame: Baseline and timepoint at which third right heart catheterization was performed, which occurred between Month 18 and Month 24
Population: All randomized participants who received their assigned treatment, transitioned to the extension period, and had data for the respective timepoints
Measure: Mean (Standard Deviation); unit: dynes*sec/cm^5
Groups:
- Placebo-Crossed Treatment Group: Participants who received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) were re-randomized to receive either 0.3 mg/kg or 0.7 mg/kg of sotatercept plus SOC during 30-month extension period (Cycles 9-51). Per protocol, for Delayed-Start Analysis, the Placebo-Crossed Treatment Group included all participants who received 0.3 mg/kg plus SOC or 0.7 mg/kg of sotatercept plus SOC after a full course of placebo, regardless of their dose level. Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Continued Sotatercept Treatment Group: Participants who were randomized to receive either 0.3 mg/kg or 0.7 mg/kg of sotatercept plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) continued to receive sotatercept 0.3 mg/kg or 0.7 mg/kg plus SOC during the 30-month extension period (Cycles 9-51). Per protocol, for Delayed-Start Analysis, the Continued Sotatercept Treatment Group combined participants who received 0.3 mg/kg or 0.7 mg/kg of sotatercept plus SOC. Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Placebo-Crossed Treatment Group | Continued Sotatercept Treatment Group
Number analyzed (Participants) | 30 | 67
dynes*sec/cm^5
  Extension Period: Change from Baseline in PVR (Delayed-Start Analysis): number analyzed (Participants) | 25 | 57
  Extension Period: Change from Baseline in PVR (Delayed-Start Analysis) | -246.9 (300.01) | -212.6 (254.24)
  Baseline | 802.0 (331.05) | 783.7 (371.59)
Statistical Analysis 1: Comparison: Placebo-Crossed Treatment Group vs Continued Sotatercept Treatment Group; Analysis based on calculated LS means; Test type: Superiority; p = 0.7851, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Squares Means = -13.9, 95% CI 2-sided [-113.85 to 86.06], Standard Error of Mean 50.95

3. Primary Outcome: Extension Period: Change From Baseline in PVR (Placebo-Crossed Analysis)
Description: as for outcome 2
Time Frame: Baseline and the timepoint at which the third right heart catheterization was performed, which occurred between Month 18 and Month 24.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dynes*sec/cm^5
Groups:
- Placebo-Crossed Treatment Group: Participants who received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) were re-randomized to receive either 0.3 mg/kg or 0.7 mg/kg of sotatercept plus SOC during 30-month extension period (Cycles 9-51). Per protocol, for Placebo-Crossed Analysis, the Placebo-Crossed Treatment Group included all participants who received 0.3 mg/kg plus SOC or 0.7 mg/kg of sotatercept plus SOC after a full course of placebo, regardless of their dose level. Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Placebo-Crossed Treatment Group
Number analyzed (Participants) | 30
dynes*sec/cm^5
  Extension Period: Change from Baseline in PVR (Placebo-Crossed Analysis): number analyzed (Participants) | 25
  Extension Period: Change from Baseline in PVR (Placebo-Crossed Analysis) | -246.9 (300.01)
  Baseline | 802.0 (331.05)
Statistical Analysis 1: Comparison: Placebo-Crossed Treatment Group; Test type: Superiority; p < .0001, ANCOVA — Comparison of baseline and final value; Multiple Imputation Mean Difference = -223.2, 95% CI 2-sided [-335.83 to -110.49], Standard Error of Mean 57.45 — Standard multiple imputations are done with imputed values that are within the range of the minimum and maximum observed values using linear regression including baseline measurements

4. Primary Outcome: Extension Period: Number of Participants Who Experienced One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a study participant administered a pharmaceutical product that does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Time Frame: Up to approximately 32 months
Population: All randomized participants who transitioned to the extension period and received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- Extension Period: Placebo→Sotatercept 0.3 mg/kg: This treatment group represents participants from the Placebo arm who received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8), then transitioned to the 30-month extension period (Cycles 9-51), during which they received sotatercept 0.3 mg/kg plus SOC by SC injection. Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Extension Period: Sotatercept 0.3 mg/kg: Participants who received sotatercept 0.3 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) continued to receive sotatercept 0.3 mg/kg plus SOC during the 30-month extension period (Cycles 9-51). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Extension Period: Sotatercept 0.7 mg/kg: Participants who received sotatercept 0.7 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8) continued to receive sotatercept 0.7 mg/kg plus SOC during the 30-month extension period (Cycles 9-51). Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Extension Period: Placebo→Sotatercept 0.3 mg/kg | Extension Period: Placebo→Sotatercept 0.7 mg/kg | Extension Period: Sotatercept 0.3 mg/kg | Extension Period: Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 15 | 15 | 31 | 36
Participants | 14 | 15 | 31 | 36

5. Primary Outcome: Extension Period: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to 30 months
Population: All randomized participants who transitioned to the extension period and received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Extension Period: Placebo→Sotatercept 0.3 mg/kg | Extension Period: Placebo→Sotatercept 0.7 mg/kg | Extension Period: Sotatercept 0.3 mg/kg | Extension Period: Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 15 | 15 | 31 | 36
Participants | 1 | 0 | 1 | 3

6. Secondary Outcome: Base Study: Change From Baseline in 6-Minute Walk Distance (6MWD) at 24 Weeks
Description: 6MWD is measured by an exercise test known as 6-Minute Walk Test (6MWT) that assesses aerobic capacity and endurance. It measures the distance covered over a time of 6 minutes and is used as an outcome measure by which to compare changes in performance capacity. Each participant's 6MWD was measured at baseline and at 24 weeks. An increase in the distance walked during the 6MWT indicates improvement in basic mobility.
Time Frame: Baseline and 24 weeks
Population: All randomized participants administered their assigned treatment who received at least 6 of the same doses during Base Study, had baseline and post-Base Study PVR assessment and EOT assessment. Note: Data from participants whose dose was down-titrated were analyzed according to dose received at least 6 times rather than dose originally assigned. Per protocol, only participants who consistently received in 0.3 mg/kg or 0.7 mg/kg of sotatercept were planned to be analyzed.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 27 | 30
meters | 31.4 (9.69) | 56.0 (10.07) | 53.6 (9.84)

7. Secondary Outcome: Base Study: Change From Baseline in Concentration of Amino-Terminal Brain Natriuretic Propeptide (NT-proBNP) at 24 Weeks
Description: Each participant's laboratory biomarkers N-terminal prohormone brain-type natriuretic peptide (NT-proBNP) or brain-type natriuretic peptide (BNP) were measured at baseline and at 24 weeks.
Time Frame: Baseline and 24 Weeks
Population: All randomized participants administered their assigned treatment who received ≥6 of the same doses during Base Study, had baseline and post-Base Study PVR assessment and EOT assessment, and had data for the outcome measure. Note: Data from participants whose dose was down-titrated were analyzed according to dose received ≥6 times rather than dose originally assigned. Per protocol, only participants who consistently received in 0.3 mg/kg or 0.7 mg/kg of sotatercept were planned to be analyzed.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 29 | 25 | 28
pg/mL | 195.9 (726.46) | -718.2 (965.12) | -359.0 (757.58)

8. Secondary Outcome: Base Study: Change From Baseline in Tricuspid Annular Plane Systolic Excursion (TAPSE) at 24 Weeks
Description: Each participant's TAPSE, which is commonly used to evaluate tricuspid valve annulus movement as an indicator of right heart function, was measured by echocardiography at baseline and 24 weeks.
Time Frame: Baseline and 24 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 28 | 24 | 28
cm | 0.0 (0.39) | 0.1 (0.26) | -0.1 (0.34)

9. Secondary Outcome: Base Study: Change From Baseline in Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) Score at Cycle 9
Description: The CAMPHOR is participant-reported questionnaire that contains 65 items in total, 25 relating to symptoms, 25 relating to quality of life (QoL), and 15 relating to activities. Symptom items are scored from 0-25, with a higher score indicating worse symptoms. QoL items are also scored from 0-25, with a higher score indicating a worse QoL and greater functional limitation. Activity items are scored from 0-30, with a higher score indicating poorer functioning. The combined score is obtained by summing up the symptoms score, QoL score and activity score. The lowest combined score possible is 0, while the highest combined score possible is 80. Each participant's CAMPHOR score was recorded at baseline and on Day 1 of Cycle 9.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 29 | 23 | 21
Score on a scale | -10.2 (12.91) | -6.9 (12.51) | -7.5 (7.96)

10. Secondary Outcome: Base Study: Change From Baseline in 36-Item Short Form Health Survey (SF-36) Score
Description: The SF-36 questionnaire is a participant-reported survey of a participant's health. The survey evaluates 8 aspects of functional health and well-being that relate to either physical health or mental health. The physical component summary is based primarily on physical functioning, bodily pain, and general health. The mental component summary encompasses vitality, social functioning, and emotional and mental health. Total scores for the physical component range from 0-100, with 100 representing the highest level of physical functioning. The total scores for the mental component also range from 0-100, with 100 representing the highest level of mental functioning. Each participant's SF-36 was recorded at baseline and on Day 1 of Cycle 9. Each cycle was 21 days.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 27 | 29
Score on a scale
  Physical component | 3.5 (1.07) | 4.5 (1.12) | 3.1 (1.11)
  Mental component | 3.2 (1.33) | 3.6 (1.39) | 0.0 (1.40)

11. Secondary Outcome: Base Study: Number of Participants Who Experienced Events Indicative of Clinical Worsening of Pulmonary Arterial Hypertension (PAH)
Description: Events that indicate clinical worsening of PAH include death, need for and/or worsening-related listing for lung and/or heart transplant, need to initiate an approved PAH SOC rescue therapy, PAH-specific hospitalization, or functional deterioration (worsened WHO Functional Class AND 15% decrease in 6MWD).
Time Frame: Up to 24 weeks
Population: All randomized participants who received their assigned treatment and had data for Base Study: Number of Participants Who Experienced Events Indicative of Clinical Worsening of PAH
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 32 | 32 | 42
Participants | 2 | 0 | 1

12. Secondary Outcome: Base Study: Number of Participants Who Experienced an Improvement From Baseline in World Health Organization (WHO) Functional Class at 24 Weeks
Description: The WHO Functional Class describes the severity of a person's pulmonary hypertension symptoms. There are four different classes: I is the mildest and IV the most severe form of pulmonary hypertension.
Time Frame: Baseline and 24 Weeks
Population: All randomized participants who received their assigned treatment and at least 6 of the same doses during Base Study, had baseline and post-Base Study PVR assessment and EOT assessment, and had data for Base Study: Number of Participants Who Experienced an Improvement from Baseline in WHO Functional Class at 24 Weeks. Note: Data from participants whose dose was down-titrated were analyzed according to dose received at least 6 times rather than dose to which originally assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 27 | 30
Participants | 4 | 8 | 6

13. Secondary Outcome: Base Study: Number of Participants Who Experienced One or More AEs
Description: as for outcome 4
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 32 | 32 | 42
Participants | 29 | 29 | 35

14. Secondary Outcome: Base Study: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to 24 weeks
Population: All randomized participants who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 32 | 32 | 42
Participants | 1 | 1 | 5

15. Secondary Outcome: Base Study: Change From Baseline in Body Mass Index (BMI) at Cycle 9
Description: Each participant's BMI was measured at baseline and at 24 weeks.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: All randomized participants who received their assigned treatment and had data for Base Study: Change from Baseline in BMI at Cycle 9
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 31 | 36
kg/m^2 | -0.2 (1.25) | 0.6 (0.89) | 0.2 (1.07)

16. Secondary Outcome: Base Study: Change From Baseline in Systolic and Diastolic Blood Pressure at Cycle 9
Description: Each participant's systolic and diastolic blood pressure was taken at baseline and on Day 1 of Cycle 9. Each cycle was 21 days.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: All randomized participants who received their assigned treatment and had data for Base Study: Change from Baseline in Systolic and Diastolic Blood Pressure at Cycle 9
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 31 | 36
mmHg
  Systolic blood pressure | -0.8 (10.06) | 3.4 (11.75) | 2.6 (12.28)
  Diastolic blood pressure | 2.3 (8.06) | 4.1 (8.64) | 1.7 (8.69)

17. Secondary Outcome: Base Study: Change From Baseline in Respiratory Rate at Cycle 9
Description: Each participant's respiratory rate (number of breaths per minute) was measured at baseline and on Day 1 of Cycle 9. Each cycle was 21 days.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: All randomized participants who received their assigned treatment and had data for Base Study: Change from Baseline in Respiratory Rate at Cycle 9
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 29 | 31 | 36
breaths/min | -0.3 (2.10) | -1.3 (3.72) | -0.3 (3.05)

18. Secondary Outcome: Base Study: Change From Baseline in QTcF Interval at Cycle 9
Description: Each participant's QTcF Interval was measured at baseline and on Day 1 of Cycle 9.
Time Frame: Baseline and Day 1 of Cycle 9, up to 24 weeks (Each cycle was 21 days.)
Population: All randomized participants who received their assigned treatment and had data for Base Study: Change from Baseline in QTcF Interval at Cycle 9
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Placebo | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 30 | 31 | 35
milliseconds | 0.7 (31.10) | -7.4 (20.57) | -9.1 (31.55)

19. Secondary Outcome: Base Study: Maximum Plasma Concentration (Cmax) of Sotatercept
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose is given. Based on population pharmacokinetic (PopPK) modeling of previous sotatercept studies, Cmax occurs at Day 8 of Cycle 1 after a sotatercept dose is given. The sotatercept concentration at Day 8 of Cycle 1 (each cycle was 21 days) is presented here as Cmax.
Time Frame: Day 8 of Cycle 1 (Each cycle was 21 days.)
Population: All randomized participants who received at least 1 dose of sotatercept and had sufficient pharmacokinetic samples collected and assayed for PK analysis
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Sotatercept 0.3 mg/kg: Participants received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Sotatercept 0.3 mg/kg | Sotatercept 0.7 mg/kg
Number analyzed (Participants) | 32 | 42
ng/mL | 1910.3 (715.86) | 4598.5 (1622.59)

20. Secondary Outcome: Extension Period: Change From Baseline in 6MWD (Delayed-Start Analysis)
Description: 6MWD is measured by an exercise test known as 6MWT that assesses aerobic capacity and endurance. It measures the distance covered over a time of 6 minutes and is used as an outcome measure by which to compare changes in performance capacity. Each participant's 6MWD was measured at baseline and the timepoint at which the third RCH was performed. This occurred between Month 18 and Month 24, at which time each participant's 6MWD was also measured. An increase in the distance walked during the 6MWT indicates improvement in basic mobility.
Time Frame: Baseline and the timepoint at which third right heart catheterization was performed, which occurred between Month 18 and Month 24
Population: All randomized participants who received their assigned treatment, transitioned to the extension period, and had data for Extension Period: Change from Baseline in 6MWD (Delayed-Start Analysis)
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo-Crossed Treatment Group | Continued Sotatercept Treatment Group
Number analyzed (Participants) | 30 | 67
meters | 60.1 (14.35) | 55.7 (9.47)

21. Secondary Outcome: Extension Period: Change From Baseline in 6MWD (Placebo-Crossed Analysis)
Description: 6MWD is measured by an exercise test known as 6MWT that assesses aerobic capacity and endurance. It measures the distance covered over a time of 6 minutes and is used as an outcome measure by which to compare changes in performance capacity. Each participant's 6MWD was measured at baseline and the timepoint at which the third right heart catheterization was performed. This occurred between Month 18 and Month 24, at which time each participant's 6MWD was also measured. An increase in the distance walked during the 6MWT indicates improvement in basic mobility.
Time Frame: as for outcome 2
Population: All randomized participants who received their assigned treatment, transitioned to the extension period, and had data for Extension Period: Change from Baseline in 6MWD (Placebo-Crossed Analysis)
Measure: Mean (Standard Error); unit: meters
Arm/Group | Placebo-Crossed Treatment Group
Number analyzed (Participants) | 30
meters | 60.5 (13.21)

22. Secondary Outcome: Extension Period: Number of Participants Who Experienced an Improvement From Baseline in WHO Functional Class (Delayed-Start Analysis)
Description: The WHO Functional Class describes the severity of a person's pulmonary hypertension symptoms. There are four different classes: I is the mildest and IV the most severe form of pulmonary hypertension. Each participant's WHO Functional Class was assessed at baseline and the timepoint at which the third right heart catheterization was performed. This occurred between Month 18 and Month 24, at which time each participant's WHO Functional Class was also assessed.
Time Frame: as for outcome 2
Population: All randomized participants who received their assigned treatment, transitioned to the extension period, and had data for Extension Period: Number of Participants Who Experienced an Improvement from Baseline in WHO Functional Class (Delayed-Start Analysis)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo-Crossed Treatment Group | Continued Sotatercept Treatment Group
Number analyzed (Participants) | 29 | 66
Participants | 16 | 27

23. Secondary Outcome: Extension Period: Change From Baseline in WHO Functional Class (Placebo-Crossed Analysis)
Description: as for outcome 22
Time Frame: as for outcome 2
Population: All randomized participants who received their assigned treatment, transitioned to the extension period, and had data for Extension Period: Change from Baseline in WHO Functional Class (Placebo-Crossed Analysis)
Measure: Mean (Standard Deviation); unit: WHO functional class
Arm/Group | Placebo-Crossed Treatment Group
Number analyzed (Participants) | 28
WHO functional class | -0.6 (0.74)

ADVERSE EVENTS:
Time Frame: Treatment period: Up to 24 weeks; Extension period: Up to approximately 32 months.
Description: The safety analysis population included all participants who received at least 1 dose of study treatment. The analysis population for All-Cause Mortality included all randomized participants.
Groups:
- Base Study: Placebo: Participants received placebo plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Base Study: Sotatercept 0.3 mg/kg: Participants received sotatercept 0.3 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
- Base Study: Sotatercept 0.7 mg/kg: Participants received sotatercept 0.7 mg/kg plus SOC by SC injection during the 24-week treatment period (Base Study; Cycles 1-8). Each cycle was 21 days. Dosing occurred once every 3 weeks.
Arm/Group | Base Study: Placebo | Base Study: Sotatercept 0.3 mg/kg | Base Study: Sotatercept 0.7 mg/kg | Extension Period: Placebo→Sotatercept 0.3 mg/kg | Extension Period: Placebo→Sotatercept 0.7 mg/kg | Extension Period: Sotatercept 0.3 mg/kg | Extension Period: Sotatercept 0.7 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 1/42 | 1/15 | 0/15 | 1/32 | 2/42
Serious Adverse Events (participants affected / at risk) | 3/32 | 2/32 | 10/42 | 6/15 | 4/15 | 10/31 | 12/36
Other Adverse Events (participants affected / at risk) | 25/32 | 29/32 | 33/42 | 14/15 | 15/15 | 30/31 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Placebo (N=32) | Base Study: Sotatercept 0.3 mg/kg (N=32) | Base Study: Sotatercept 0.7 mg/kg (N=42) | Extension Period: Placebo→Sotatercept 0.3 mg/kg (N=15) | Extension Period: Placebo→Sotatercept 0.7 mg/kg (N=15) | Extension Period: Sotatercept 0.3 mg/kg (N=31) | Extension Period: Sotatercept 0.7 mg/kg (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Right ventricular failure (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Septic embolus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Base Study: Placebo (N=32) | Base Study: Sotatercept 0.3 mg/kg (N=32) | Base Study: Sotatercept 0.7 mg/kg (N=42) | Extension Period: Placebo→Sotatercept 0.3 mg/kg (N=15) | Extension Period: Placebo→Sotatercept 0.7 mg/kg (N=15) | Extension Period: Sotatercept 0.3 mg/kg (N=31) | Extension Period: Sotatercept 0.7 mg/kg (N=36)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 8 (13) | 1 (2)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 1 (1) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 5 (8) | 3 (3) | 1 (2) | 3 (3) | 3 (8)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 2 (4) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tachycardia paroxysmal (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deposit eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dental plaque (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (6) | 7 (8) | 6 (6) | 3 (3) | 5 (7) | 9 (14) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 2 (2) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (9) | 3 (4) | 5 (5) | 3 (3) | 4 (9) | 9 (11) | 5 (7)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (10) | 3 (3) | 3 (3) | 1 (3) | 3 (4) | 6 (9) | 4 (5)
Application site pain (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 2 (2)
Catheter site haemorrhage (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (6) | 2 (2) | 4 (4) | 6 (7) | 4 (5) | 6 (9) | 5 (6)
Feeling abnormal (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (4) | 2 (2)
Oedema peripheral (General disorders) | 5 (5) | 3 (3) | 5 (6) | 4 (4) | 6 (6) | 11 (12) | 7 (8)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 5 (5) | 3 (3)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder polyp (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 5 (6)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Fungal pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 2 (3) | 4 (4) | 2 (2) | 2 (2) | 5 (5) | 2 (2)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5)
Labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 4 (4) | 5 (9) | 6 (7) | 10 (14) | 1 (1)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 2 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (5) | 2 (3) | 3 (4)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 4 (5) | 2 (2) | 3 (3) | 1 (1) | 6 (9) | 6 (8)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 5 (7) | 5 (5)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 5 (5) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (4) | 2 (2) | 3 (5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood chloride increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 1 (1) | 7 (7) | 1 (1) | 5 (7) | 0 (0) | 5 (5)
Intraocular pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reticulocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Urine albumin/creatinine ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fluid retention (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 2 (6) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 5 (5) | 3 (5) | 0 (0) | 4 (8) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (6) | 2 (2) | 3 (3) | 6 (8)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1) | 2 (2) | 5 (9) | 8 (12) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 7 (10) | 2 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 4 (4) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (4) | 5 (6) | 2 (6) | 3 (3) | 8 (11) | 3 (4)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 3 (4) | 5 (5) | 4 (5) | 4 (5) | 2 (2) | 4 (6) | 5 (6)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (10) | 8 (16) | 6 (8) | 4 (21) | 7 (13) | 9 (16) | 6 (10)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intention tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (3) | 2 (3) | 2 (2) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Procedural anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (4) | 3 (4) | 4 (4) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (2) | 0 (0) | 3 (4) | 3 (6) | 5 (8) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 5 (6) | 3 (7) | 4 (5) | 7 (10) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (5) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 3 (4) | 2 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 1 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (6) | 5 (5) | 7 (8)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 3 (4)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 4 (4) | 3 (3)
Hypotension (Vascular disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 2 (12) | 2 (2) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will comply with the requirements for publication of study results. In accordance with standard editorial and ethical practice, the sponsor will generally support publication.

DOCUMENTS (2):
  • Study Protocol (2020-07-31): https://cdn.clinicaltrials.gov/large-docs/07/NCT03496207/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT03496207/SAP_001.pdf